CLINICAL TRIAL: NCT00050518
Title: A Multicenter, Double-Blind, Randomized Study of the Safety and Efficacy of Aventis Pasteur's Smallpox Vaccine, USP (APSV) in Vaccinia-Naive Adults.
Brief Title: APSV in Vaccinia Naive Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 02-054
Record Dates: First submitted 2002-12-11; First posted 2002-12-13 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-03

CONDITIONS: Smallpox
Keywords: Smallpox; Aventis Pasteur; Vaccine
MeSH Terms: conditions — Smallpox | interventions — Aventis Pasteur smallpox vaccine

INTERVENTIONS:
Biological: Aventis Pasteur Smallpox Vaccine

SUMMARY:
The study seeks to define, with precision, the safety and efficacy of APSV, two dose potencies of one lot in vaccinia-naive adults. The ability of this vaccine to induce a classic �take� as defined by formation of a lesion at the injection site consistent with the �Jennerian� process (see Appendix A) and vaccine specific immune responses will be assessed. The local cutaneous lesion is considered to be a surrogate for clinical effectiveness of live, replicating smallpox vaccines. Neutralizing antibody formation has been correlated with takes for the Dryvax vaccine and is considered to be cross-protective for other orthopoxviruses, including variola. The study also seeks to characterize preliminarily the cell mediated immune (CMI) response to APSV (as compared to Dryvax).

DETAILED DESCRIPTION:
A Multicenter, double blind, randomized trial in which each volunteer will receive one of 2 dose concentrations of one of two lots of Aventis Pasteur Smallpox Vaccine as a single vaccination (undiluted, 1:5 dilution). Volunteers without a take at day 7 - 9 will be offered a vaccination with Dryvax at the end of the study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Adequate renal function defined as a serum creatinine 1.5 mg/dL; urine protein < 100mg/ dL or trace or negative proteinuria (by dipstick), and a calculated creatinine clearance >55 mL/min. Formula for calculations is contained within the Manual of Procedures.

(Note: Renal function is measured to ensure that subjects could meet criteria for use of cidofovir if needed).

* Age 18-32 (children are excluded due to concerns of safety, including autoinoculation).
* Willing to sign informed consent.
* Availability for follow-up for planned duration of the study (56 days following the last vaccination).
* Acceptable medical history by screen evaluation form and brief assessment.
* Absence of a typical vaccinia scar and negative history of smallpox vaccination.
* Negative urine or serum pregnancy test for women of childbearing potential.
* If the volunteer is female and of childbearing potential, she agrees to use acceptable contraception, and not become pregnant for the duration of the study. (Acceptable contraception includes implants, injectables, combined oral contraceptives, effective intrauterine devices (IUDs), sexual abstinence, or a vasectomized partner).
* Negative ELISA for HIV or negative Western blot for subjects who have a positive ELISA and have participated in an HIV vaccine trial.
* Negative hepatitis B surface antigen and negative antibody to hepatitis C virus.
* Negative urine glucose by dipstick.
* ALT < 1.5 times institutional upper limit of normal.

EXCLUSION CRITERIA:

* Allergies to any component of the vaccines (e.g., polymyxin B sulfate, dihydrostreptomycin sulfate, chlorotetracycline hydrochloride).
* History of immunodeficiency.
* Serology positive for HIV, hepatitis B, or hepatitis C at the screening visit.
* Known or suspected impairment of immunologic function including, but not limited to clinically significant liver disease.
* Diabetes mellitus.
* Moderate to severe kidney impairment.
* Malignancy with the exception of squamous cell or basal cell skin cancer.
* Autoimmune disease.
* Use of immunosuppressive medication.
* Corticosteroid nasal sprays are permissible.
* Medical or psychiatric condition or occupational responsibilities which preclude subject compliance with the protocol.
* History of illegal injection drug use.
* Live attenuated vaccines within 60 days of study.
* Use of experimental agents within 30 days prior to study.
* Any history of vaccination with any vaccinia vectored or other pox vectored experimental vaccine.
* Smallpox vaccination since 1990 (Vaccinia experience cohorts).
* Typical vaccinia scar or history of smallpox vaccination (Vaccinia naive cohorts only).
* Receipt of blood products or immunoglobulin in the past 6 months.
* Recent donation of the equivalent of a pint of blood within the 30 days prior to enrollment.
* Acute febrile illness (100.5 F) on the day of vaccination.
* Pregnant or lactating women.
* Eczema of any degree or history of eczema.
* History of exfoliative skin disorders/conditions.
* Any acute skin disorders of large magnitude, e.g., laceration requiring sutures, burn greater than 2x2 cm.
* Household contacts/sexual contacts with, or close and frequent occupational exposure to, any of the following: pregnant women, children < 12 months of age, people with eczema or history of eczema, people with any of the skin disorders/conditions previously listed, people with immunodeficiency disease or use of immunosuppressive medications.
* Any condition which, in the opinion of the investigator, might interfere with study objectives.

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 444
Dates: Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Iowa - Iowa City IA, Iowa City, Iowa
  - Cincinnati Children's Hospital Med Ctr, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Vanderbilt University, Nashville, Tennessee